CLINICAL TRIAL: NCT02376374
Title: OPV Transmissibility in Communities After Cessation of Routine OPV Immunization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Instituto Nacional de Salud Publica, Mexico (Other)
Responsible Party: Principal Investigator, Yvonne (Bonnie) A Maldonado, OPV transmissibility in communities after cessation of routine OPV immunization, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 31546
Record Dates: First submitted 2015-02-18; First posted 2015-03-03 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Polio
Keywords: transmission; vaccine
MeSH Terms: conditions — Poliomyelitis | interventions — Residence Characteristics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 10% OPV (Experimental): In this arm, 10% of the households in this community will receive OPV.
  Interventions: Other: Controlling vaccination rates in communities
- 30% OPV (Experimental): In this arm, 30% of the households in this community will receive OPV.
  Interventions: Other: Controlling vaccination rates in communities
- 70% OPV (Experimental): In this arm, 70% of the households in this community will receive OPV.
  Interventions: Other: Controlling vaccination rates in communities

INTERVENTIONS:
Other: Controlling vaccination rates in communities — Three communities will be in three arms, one per arm. From 150 randomly-selected households, 10% will receive OPV in one community, 30% in the second community, and 70% in the third community.

SUMMARY:
The investigators propose to study both inter- and intra-household Oral Polio Vaccine (OPV) transmission in a primarily inactivated-polio vaccine (IPV)-vaccinated community in Mexico. The investigators will enroll 3 distinct clusters of households in a municipality in Orizaba, Veracruz, Mexico prior to the February 2015 National Immunization Week (NIW.) These clusters will be physically separate from one another and differ only in the proportion of OPV-eligible children who will receive OPV during the February 2015 NIW (10%, 30% and 70% vaccinated.) The investigators will look at inter-household and intra-household transmission. The investigators will then determine if epidemiologic (i.e.: degree of contact), anthropometric (i.e.: nutritional status) or clinical covariates (i.e.: IPV/OPV immunization history) are associated with intra-household transmission.

DETAILED DESCRIPTION:
We propose a prospective study to be conducted in 3 distinct clusters of 150 households each in one semi-urban municipality in Orizaba, Veracruz, Mexico during and after the February 2015 National Immunization Week (NIW.) Mexico provides a unique environment to study OPV transmission. The last case of poliomyelitis was reported in 1990. Mexico transitioned from an OPV to an IPV-based immunization regimen in 2007-2008. Currently, Mexican children receive IPV at 2, 4, 6, and 18 months of age. In addition, children ≤5 years old who have received at least 2 doses of IPV are eligible to receive OPV during biannual NIW held in February and May each year. Because of the changes in vaccination regimens over time, Mexican households consist of individuals with different degrees of susceptibility to OPV infection: those born before 2007 who were exposed to WPV and OPV or OPV alone, those born after 2007 exposed to IPV with intermittent OPV exposure, and un-vaccinated infants, some with maternal polio virus antibodies. By studying OPV transmission in this setting, we will be able to assess the impact of differing immunization status on OPV shedding and transmission.

We will conduct our study in a relatively isolated and semi-urban municipality of Orizaba, Veracruz, Mexico. These household clusters will differ only in the proportion of OPV-eligible children who will be OPV-vaccinated during the February 2015 National Immunization Week (10%, 30% and 70%.) We will enroll households that have at least 1 healthy child less than 5 years of age with an up-to-date IPV vaccination history. Enrolled households will then be randomized to the OPV-vaccinated or non-vaccinated arm of each household cluster. Eligible children from households in the OPV-vaccinated arm will then be further randomized to either receive OPV or remain un-vaccinated. Thus, only one child per household in the OPV-vaccinated arm will be vaccinated.

We will collect stool samples from all members of the enrolled households serially over the course of the study and will determine if individuals shed OPV in their stool using a serotype-specific real-time polymerase chain reaction (PCR) assay. We will define inter-household transmission as fecal OPV shedding by any member of a non-vaccinated household. By comparing inter-household transmission rates among all the household clusters, we will determine the if the proportion of OPV-vaccinated children impacts community OPV transmission in a primarily IPV-vaccinated community. These results will be critical to predicting the risk of OPV re-introduction in the event of a poliomyelitis outbreak in the post-OPV era.

We will define intra-household transmission as OPV shedding by household contacts living in vaccinated households. We will examine intra-household transmission in all clusters together to determine if certain characteristics are associated with transmission to household contacts. Elucidating these characteristics would allow for targeted interventions to reduce or prevent OPV transmission as cessation policy is implemented or in the event that OPV re-introduction is needed during polio endgame.

ELIGIBILITY:
Inclusion Criteria:

* Households with children under the age of 5 who have up-to-date IPV vaccination history and willing to give informed consent and/or assent.

Exclusion Criteria:

* Unwilling/unable to bring children's IPV vaccination records up-to-date.

Max Age: 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1828 (Actual)
Dates: Start 2015-02; Primary Completion 2017-02-28 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Inter-household transmission of poliovirus | Feb 2015-May 2015; 4 months
Intra-household transmission of poliovirus | Feb 2015-May 2015; 4 months

DOCUMENTS (1):
  • Study Protocol (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/74/NCT02376374/Prot_000.pdf